CLINICAL TRIAL: NCT06615765
Title: Efficacy and Safety of Two-step Acupuncture Therapy for Symptom Relief in Adults with Mild to Moderate Ulcerative Colitis
Brief Title: Acupuncture for Symptom Relief in Adults with Mild to Moderate Ulcerative Colitis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guang'anmen Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, He Chen, Researcher, Department of Acupuncture, Guang'anmen Hospital, China Academy of Chinese Medical Sciences, Principal Investigator, Guang'anmen Hospital of China Academy of Chinese Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-190-KY
Record Dates: First submitted 2024-09-22; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Ulcerative Colitis
Keywords: Acupuncture; Ulcerative colitis; Patient-reported outcome 2; Inflammatory bowel disease; Randomized controlled trial
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding will be maintained for participants, outcome assessors, and statisticians to prevent bias in evaluation. However, the practitioner administering the intervention will not be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acupuncture group (Experimental): Acupuncture sessions will use sterile, disposable stainless-steel needles (0.3 mm × 40 mm and 0.3 mm × 75 mm). Each session has two phases:
  Supine Position:
  Needles (0.35 mm × 75 mm) are inserted into ST25, ST15, and SP14, reaching the abdominal muscle layer.
  Needles (0.30 mm × 40 mm) are inserted into CV12, CV4, ST36, ST37, and SP6. Electroacupuncture (EA) at ST25, SP15, and ST36 uses a continuous 5 Hz wave, 0.1 to 2.0 mA.
  Prone Position:
  Needles are inserted into BL32, BL33, and BL35 with precise angles and depths. EA at BL32, BL33, and BL35 uses a continuous 5 Hz wave, 2.0 to 6.5 mA. Sessions occur three times a week for the first 4 weeks, then twice a week for weeks 5 to 8, each lasting 40 minutes, totaling 20 sessions.
  Interventions: Other: Acupuncture
- Sham acupuncture group (Sham Comparator): Sterile, disposable stainless-steel needles (0.30 mm × 25 mm) will be used. After skin sterilization, needles will be inserted into the same points as the acupuncture group but to a shallow depth of 2 to 3 mm and lightly manipulated for blinding. Paired alligator clips will be attached to the same points, but the sham EA apparatus will have no current output, though it mimics the active EA apparatus in appearance and sound. Sham sessions will follow the same schedule as the acupuncture group: three times a week for the first 4 weeks and twice a week for weeks 5 to 8, each lasting 40 minutes, totaling 20 sessions.
  Interventions: Other: Sham acupuncture

INTERVENTIONS:
Other: Acupuncture — Acupuncture sessions will use sterile, disposable stainless-steel needles (0.3 mm × 40 mm and 0.3 mm × 75 mm). Each session has two phases:
  Supine Position:
  * Needles (0.35 mm × 75 mm) are inserted into ST25, ST15, and SP14, reaching the abdominal muscle layer.
  * Needles (0.30 mm × 40 mm) are inserted into CV12, CV4, ST36, ST37, and SP6.
  * Electroacupuncture (EA) at ST25, SP15, and ST36 uses a continuous 5 Hz wave, 0.1 to 2.0 mA.
  Prone Position:
  * Needles are inserted into BL32, BL33, and BL35 with precise angles and depths.
  * EA at BL32, BL33, and BL35 uses a continuous 5 Hz wave, 2.0 to 6.5 mA. Sessions occur three times a week for the first 4 weeks, then twice a week for weeks 5 to 8, each lasting 40 minutes, totaling 20 sessions.
  Arms: Acupuncture group
Other: Sham acupuncture — Sterile, disposable stainless-steel needles (0.30 mm × 25 mm) will be used. After skin sterilization, needles will be inserted into the same points as the acupuncture group but to a shallow depth of 2 to 3 mm and lightly manipulated for blinding. Paired alligator clips will be attached to the same points, but the sham EA apparatus will have no current output, though it mimics the active EA apparatus in appearance and sound. Sham sessions will follow the same schedule as the acupuncture group: three times a week for the first 4 weeks and twice a week for weeks 5 to 8, each lasting 40 minutes, totaling 20 sessions.
  Arms: Sham acupuncture group

SUMMARY:
Ulcerative colitis (UC) is one of the two primary forms of inflammatory bowel disease. This condition is characterized by continuous mucosal inflammation that begins in the rectum and extends proximally throughout the colon. Common intestinal symptoms also include rectal bleeding, increased stool frequency, tenesmus, nocturnal bowel movements, and crampy abdominal pain. Acupuncture has been suggested as a potential intervention to alleviate clinical symptoms of UC. This single-center, parallel-group, two-arm, randomized, sham-controlled trial aims to evaluate the effects and safety of acupuncture for UC.

DETAILED DESCRIPTION:
Ulcerative colitis (UC) is a chronic inflammatory bowel disease characterized by episodes of symptoms including rectal bleeding, increase stool frequency, and abdominal pain, impacting quality of life significantly. Conventional treatments often come with potential side effects and may not be sufficient. Acupuncture is increasingly recognized for its promising benefits in UC. This study aims to assess the efficacy and safety of acupuncture for symptom relief in mild to moderate UC.This single-center, parallel-arm, randomized, sham-controlled trial will involve 64 patients with UC, randomly assigned in a 1:1 ratio to either the acupuncture or sham acupuncture group. Participants will receive 20 sessions of acupuncture or sham acupuncture over eight weeks. Blinding will be applied to participants, outcome assessors, and statisticians. The primary outcome measure is the change in Patient-Reported Outcome 2 (PRO2) from baseline at week 8. Secondary outcomes include changes from baseline in the following scales: PRO2 at other time points, weekly average Numeric Rating Scale (U-NRS) for bowel urgency, weekly average NRS for abdominal pain (both associated and not associated with bowel movement), the 32-item Inflammatory Bowel Disease Questionnaire (IBDQ-32), Work Productivity and Activity Impairment Questionnaire-Inflammatory Bowel Disease (WPAI-IBD), Pittsburgh Sleep Quality Index (PSQI), and Hospital Anxiety and Depression Scale (HADS). Patient Global Impression of Change (PGIC) will also be assessed as secondary outcomes. Adverse events and additional treatments will be monitored throughout the study. The modified intention-to-treat (mITT) population will include participants who complete baseline assessments and receive at least one treatment session.

ELIGIBILITY:
Inclusion Criteria:

Eligible participants are those aged 18 to 70 years who meet the diagnostic criteria for mild to moderate UC, have a PRO2 score of ≥ 2 points, and provide written informed consent. Patients currently receiving oral and/or topical 5-aminosalicylic acid (such as mesalamine) may continue their treatment during the study period.

Exclusion Criteria:

Participants will be excluded if they meet any of the following criteria:

1. Diagnosis of Crohn's disease, intestinal tuberculosis, chronic intestinal infections, or intestinal malignancies.
2. Current treatment with corticosteroids, thiopurines, biologics, or oral small molecules.
3. Severe skin conditions or infections.
4. Presence of severe underlying medical conditions, including but not limited to cardiovascular diseases, hepatobiliary diseases, kidney diseases, hematologic disorders, autoimmune diseases, communicable diseases, severe malnutrition, or malignancies.
5. Mental illness, cognitive dysfunction, or language disorders.
6. Receipt of acupuncture therapy for UC within the past month.
7. Substance abuse issues.
8. Pregnancy, plans to become pregnant within the next year, lactation, or being within 12 months postpartum.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
change from baseline in the PRO2 score | Week 8 after randomization
  Data on daily bowel movements and rectal bleeding will be summarized from the stool diaries. The PRO2 score, assessed at weeks 4, 8, 12, 16, 20, 24, 28, and 32, comprises the Stool Frequency (SF) and Rectal Bleeding (RB) subscales of the Mayo score. The SF subscale is rated as follows: 0 (normal stool frequency), 1 (1-2 stools more than normal), 2 (3-4 stools more than normal), and 3 (5 or more stools more than normal). The RB subscale is rated as: 0 (no blood), 1 (streaks of blood less than half the time), 2 (obvious blood most of the time), and 3 (blood alone). The primary outcome is the change from baseline in the PRO2 score at week 8.

SECONDARY OUTCOMES:
The proportion of patients achieving a ≥ 50% reduction in PRO2 score at weeks 4, 8, 12, 16, 20, 24, 28, and 32. | Weeks 4, 8, 12, 16, 20, 24, 28, and 32 after randomization.
The proportion of patients with a PRO2 score of 0 | At weeks 4, 8, 12, 16, 20, 24, 28, and 32 after randomization.
Changes from baseline in weekly average U-NRS scores | At weeks 4, 8, 12, 16, 20, 24, 28, and 32 after randomization.
  Since bowel urgency is an independent and critical symptom impacting patients' quality of life and productivity, this study will assess bowel urgency severity using the Numeric Rating Scale (U-NRS) (0 = no urgency, 10 = worst possible urgency). The minimal clinically important difference (MCID) is defined as a ≥3-point decrease in U-NRS from baseline, while bowel urgency remission is defined as a U-NRS score of 0 or 1. In this study, patients will be instructed to record their scores for each bowel movement. The average U-NRS score will be calculated weekly by summing the U-NRS scores for the week and dividing by the total number of bowel movements.
Changes from baseline in weekly average NRS scores for abdominal pain associated with bowel movements | At weeks 4, 8, 12, 16, 20, 24, 28, and 32 after randomization.
  For the NRS score related to abdominal pain associated with bowel movements (scale 0 to 10, with higher scores indicating more severe pain), patients will record their scores for each bowel movement. The weekly average NRS score will be derived by summing these scores and dividing by the total number of bowel movements.
Changes from baseline in weekly average NRS scores for abdominal pain not associated with bowel movements | At weeks 4, 8, 12, 16, 20, 24, 28, and 32 after randomization.
  For the NRS score related to abdominal pain not associated with bowel movements (scale 0 to 10, with higher scores indicating more severe pain), patients will record daily scores, which will then be summed over the week and divided by 7 to obtain the weekly average NRS score.
Changes from baseline in IBDQ-32 scores | At weeks 4, 8, 12, 20, and 32 after randomization.
  The IBDQ-32 is the predominant tool for assessing disease-specific quality of life in randomized clinical trials for UC. Studies support the efficacy of IBDQ-32 in capturing treatment impacts on the quality of life of UC patients. The questionnaire encompasses four domains reflecting the impact of UC on patients: symptoms, psychological and social functioning, and physical and emotional well-being.
Changes from baseline in WPAI-IBD scores | At weeks 4, 8, 20, and 32 after randomization.
  The WPAI-IBD (version 2.0) (www.reillyassociates.net), is a validated tool designed to assess impairments in work and daily activities. This 6-item questionnaire evaluates impairments experienced over the past 7 days and provides four key metrics: 1) Absenteeism (percentage of work time missed); 2) Presenteeism (percentage of impairment while at work); 3) Overall work productivity loss (combined estimate of absenteeism and presenteeism); and 4) Activity impairment (percentage of impairment in daily activities). WPAI-IBD results are reported as percentages, with higher scores reflecting greater impairment and reduced productivity.
Changes from baseline in PSQI scores | At weeks 8, 20, and 32 after randomization.
  The Pittsburgh Sleep Quality Index (PSQI) is a self-administered questionnaire that assesses sleep quality and disturbances over the past month, with higher scores indicating worse sleep quality.
Changes from baseline in HADS scores | At weeks 8, 20, and 32 after randomization.
  The Hospital Anxiety and Depression Scale (HADS) is a self-report tool designed to identify symptoms of depression and anxiety, with higher scores reflecting more severe symptoms.
PGIC | At weeks 4, 8, 20, and 32 after randomization.
  The Patient Global Impression of Change (PGIC) will be used to evaluate overall improvement. This simple, patient-reported outcome measures participants' perceptions of changes in their condition using a 7-point scale: "very much improved," "much improved," "minimally improved," "no change," "minimally worse," "much worse," or "very much worse."
Changes from baseline in the PRO2 score | Weeks 4, 12, 16, 20, 24, 28, and 32 after randomization
  Data on daily bowel movements and rectal bleeding will be summarized from the stool diaries. The PRO2 score, assessed at weeks 4, 8, 12, 16, 20, 24, 28, and 32, comprises the Stool Frequency (SF) and Rectal Bleeding (RB) subscales of the Mayo score. The SF subscale is rated as follows: 0 (normal stool frequency), 1 (1-2 stools more than normal), 2 (3-4 stools more than normal), and 3 (5 or more stools more than normal). The RB subscale is rated as: 0 (no blood), 1 (streaks of blood less than half the time), 2 (obvious blood most of the time), and 3 (blood alone).

OTHER OUTCOMES:
Adverse events | Up to week 30.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chen H, Fang J, Liu S, Gao S, Shi H, Ma JZ, Shen X, Wang W, Liu Z. Efficacy and safety of two-step acupuncture therapy for symptom relief in adults with mild to moderate ulcerative colitis: rationale and design of the TSA-UC randomised controlled trial. BMJ Open. 2025 Feb 27;15(2):e094301. doi: 10.1136/bmjopen-2024-094301. PMID 40021194